CLINICAL TRIAL: NCT01356719
Title: LUNAR Study - Develop and Validate a Bedside Scoring Method for Describing the Position and Orientation of a Tracheostomy Tube Tip When Viewed Endoscopically From a Standardised Position
Brief Title: Scoring Method for Describing the Position of a Tracheostomy Tube
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: LUNAR2011
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Tracheostomy
Keywords: Tracheostomy; adverse effects; Critical Care; standards; safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tracheostomies are artificial airway devices inserted into the neck. They can become displaced and lead to patient harm. Other than external visual inspection, there is no currently described system for describing the position of a tracheostomy tube within the airway. The investigators propose to undertake endoscopic inspection of the tracheostomy tube with a small fibre-optic camera from above and also through the tube to visualise its position within the airway. The investigators will take anonymised paired images and then score these using 6 different scoring systems. The investigators will determine which scoring system provides the simplest and most reproducible scores between 6 blinded assessors. A clinically useful scoring system could be used in future to predict problems with tracheostomy positioning.

DETAILED DESCRIPTION:
Aims & Outcomes

1. Develop an appropriate bedside scoring method for describing the position and orientation of a tracheostomy tube tip when viewed endoscopically from a standardised position
2. Secondary aims

   * Correlate the endoscopic views of the tracheostomy tube with the trans-laryngeal views.
   * Is it possible to predict the trans-laryngeal view from the endoscopic view.
   * Does the position of a tracheostomy tube tip change when the patient is repositioned following percutaneous tracheostomy (when viewed endoscopically)
   * Equipment training: Compare the number of supervised endoscopies required to consistently achieve the required standardised view
3. Primary outcome

   - Determine the scoring system with the best inter-rater agreement as defined by weighted kappa and intra-class correlation coefficients.
4. Secondary outcome

   - Assess correlation between the best scoring system (chosen by above) with the translaryngeal view
5. Tertiary aim - Assessment of training: Determine the number of attempts required to obtain adequate standardised views. This will be a manikin based assessment to demonstrate competence in performing the endoscopies for the study before any procedures are undertaken on patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults >16 years old
* Presence of a percutaneous or surgical tracheostomy
* Patient being cared for in the AICU of UHSM

Exclusion Criteria:

* Endoscopy not clinically appropriate (in the opinion of the attending physician)
* Refusal by patient or their representative

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (>16yrs) who have a tracheostomy performed as part of their intensive care management
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Determine the scoring system with the best inter-rater agreement as defined by weighted kappa and intra-class correlation coefficients. | 6 months
  Determine the scoring system with the best inter-rater agreement as defined by weighted kappa and intra-class correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan A McGrath, MB ChB, Principal Investigator — University Hospital of South Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, United Kingdom

REFERENCES:
- [Derived] McGrath BA, Lynch K, Templeton R, Webster K, Simpson W, Alexander P, Columb MO. Assessment of scoring systems to describe the position of tracheostomy tubes within the airway - the lunar study. Br J Anaesth. 2017 Jan;118(1):132-138. doi: 10.1093/bja/aew336. PMID 28039250
- See also: Related Info — http://www.tracheostomy.org.uk